CLINICAL TRIAL: NCT06627426
Title: Virtual Reality for Patient Informed Consent in Neurosurgery - a Randomized Controlled Trial
Brief Title: Virtual Reality for Patient Informed Consent in Neurosurgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ko24guzman3; 2024-01819
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: VR-based Informed Consent

STUDY DESIGN:
Intervention Model Description: Randomized, open controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-based patient informed consent (Experimental): The "intervention" group will be the on receiving VR-based patient informed consent. One surgeon from the study team will be guiding the patient through their VR model and enable them to use the VR system by themselves.
  Interventions: Other: VR-based patient informed consent
- Standard of care group (No Intervention): Group that will receive standard written informed consent

INTERVENTIONS:
Other: VR-based patient informed consent — The "intervention" group will be the on receiving VR-based patient informed consent. One surgeon from the study team will be guiding the patient through their VR model first with demonstration of the technology and the model, afterwards the patient will be enabled to use the VR system by themselves. During the whole process the patient will be able to ask questions. Depending on the planned surgery, the surgical approach as well important anatomical structures will be explained.
  Arms: VR-based patient informed consent

SUMMARY:
The goal of this randomized controlled trial is to evaluate benefits of VR (virtual reality)-based patient informed consent in neurosurgery regarding subjective patient comprehension, patient-doctor relationship and anxiety.

DETAILED DESCRIPTION:
Additionally, the investigators aim to assess the cost-benefit radio as well as feasibility in a clinical routine setting. Considering the increasing patient participation in decision-making, VR could lead to better understanding of complex surgical procedures, improving the perioperative process for both, patient and surgeon, and reduce anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18 and 75
* Surgical clipping for intracranial aneurysm, resection of vascular malformations
* Craniotomy and Resection of intracranial tumors that can be segmented for VR

Exclusion Criteria:

* Visual or auditory impairment with no sufficient aid
* Patient that had VR informed consent for surgery before
* Psychiatric illness, cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of intensity of anxiety between intervention and control group | one time assessment at day 1
  Comparison of intensity of physical and cognitive anxiety symptoms will be assessed by the questionnaire Beck Anxiety Inventory (BAI). This questionnaire consists of 21 self-reported items (four-point scale).
  min score: 39 (minimal anxiety level) max score:174 (severe anxiety)
Comparison of patient doctor relationship between intervention and control group | one time assessment at day 1
  Comparison of patient doctor relationship will be assessed by PDRQ9 (patient-doctor relationship questionnaire). The questionnaire is a 9-item scale that assesses patients' perception of the relationship with the physician. Items are scored on a 5-point Likert scale ranging from 'not at all appropriate' to 'totally appropriate'. Raw sum scores range from 9 to 45, with higher scores indicating that the patient's perception of the patient-doctor relationship is more favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Westarp, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland